CLINICAL TRIAL: NCT01629225
Title: GRK4 Polymorphisms Blood Pressure Response to Candesartan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yu Changqing, Department of Cardiovascular Diseases; Institute of Cardiovascular Diseases; Daping Hospital;, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ThirdMMU
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2013-06

CONDITIONS: Essential Hypertension
Keywords: men and women; in southwestern Han Chinese
MeSH Terms: conditions — Essential Hypertension; Multiple Endocrine Neoplasia Type 1 | interventions — candesartan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- candesartan (No Intervention): All antihypertensive agents were withdrawn before the start of a 4-6 week, single-blind, after which the patients received candesartan 10 mg or 20 mg once daily as monotherapy in a single-blind fashion. The doses were doubled after 1 weeks if DBP was ≥90 mmHg.
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Candesartan — To investigate the response to candesartan among southwestern Han Chinese with essential hypertrension
  Other Names: GRK4 polymorphisms and essential hypertrension

SUMMARY:
The purpose of this study is to investigate the association between GRK4 polymorphisms and essential hypertension in southwestern Han Chinese and test whether these polymorphisms were associated with the changes in blood pressure in patients with essential hypertension treated with angiotensin II Type antagonist candesartan.

DETAILED DESCRIPTION:
All antihypertensive agents were withdrawn before the start of a 4-6 week, single-blind, after which the patients received candesartan 10 mg or 20mg once daily as monotherapy in a single-blind fashion. The doses were doubled after 1 weeks if DBP was ≥ 90 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* men and women with mild to moderate essential hypertension in southwestern Han Chinese

Exclusion Criteria:

* subjects unwilling to participate or subjects did not have all measurement required,
* subjects who were on medications, which affect blood pressure or
* whose DNA failed to amplify and 8 with errors in Mendelian segregation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The subjects with GRK4 varirants may exert different response during 4 weeks of treatment with candesartan in patients with essential hypertension | two years

CONTACTS AND LOCATIONS:
Overall Officials: Zeng Chunyu, Doctor, Study Director — TMMU
Locations (1):
- Department of Cardiology, Daping Hospital, The Third Military Medical University, Chongqing, China

REFERENCES:
- [Derived] Cai Y, Yang Y, Chen X, He D, Zhang X, Wen X, Hu J, Fu C, Qiu D, Jose PA, Zeng C, Zhou L. Circulating "LncPPARdelta" From Monocytes as a Novel Biomarker for Coronary Artery Diseases. Medicine (Baltimore). 2016 Feb;95(6):e2360. doi: 10.1097/MD.0000000000002360. PMID 26871769
- [Derived] Yang Y, Cai Y, Wu G, Chen X, Liu Y, Wang X, Yu J, Li C, Chen X, Jose PA, Zhou L, Zeng C. Plasma long non-coding RNA, CoroMarker, a novel biomarker for diagnosis of coronary artery disease. Clin Sci (Lond). 2015 Oct 1;129(8):675-85. doi: 10.1042/CS20150121. Epub 2015 Jun 11. PMID 26201019